CLINICAL TRIAL: NCT04910763
Title: Alterations to Appetite Regulation Indices in Adults With Prediabetes Following Short-Term Aerobic vs. Resistance Exercise Training
Brief Title: Prediabetes, Exercise, and Appetite Regulation
Acronym: PEAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of institutional resources to conduct project, increased cost of conducting project due to workarounds with resources not being available, and COVID-19 pausing human subjects data collection in 2020.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Tanya Halliday, Assistant Professor, PhD, RD, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000116248
Record Dates: First submitted 2021-04-19; First posted 2021-06-02 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: PreDiabetes; Appetitive Behavior
Keywords: Resistance Exercise; Pre Diabetes; Appetite
MeSH Terms: conditions — Prediabetic State; Appetitive Behavior; Glucose Intolerance | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of the two intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance Exercise (Experimental): Resistance exercise will be training all major muscle groups 2x/week (2 days upper body, 2 days lower body) at 40-50% 1 repetition max (RM; estimated from 10 RM baseline testing) for 3 sets of 10-12 reps. This equals 4x/week for the 3 week intervention period.
  Interventions: Behavioral: Resistance Exercise

INTERVENTIONS:
Behavioral: Resistance Exercise — Increasing strength and fitness and thereby influencing hormones and perceptions involved in appetite regulation.

SUMMARY:
The purpose of the study is to learn about how type of exercise influences measures of appetite regulation.

DETAILED DESCRIPTION:
The primary objective of this study is to understand the relationship between exercise modality and appetite regulation in a population with pre-diabetes. The study includes a screening visit to ensure eligibility of participants, baseline assessments, a resistance exercise intervention, and post intervention measurements. The variables of interest include, but are not limited to, hormonal responses to exercise training pertaining to appetite, food cravings, appetite ratings. activity levels, body composition, and ten repetition-max strength. The aim of this study is to better understand the mechanisms involved in the correlation or causation of any improvements in fitness and appetite regulation in a cohort with pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years of age
* BMI between 27-40 kg/m²
* Hemoglobin A1c level between 5.7% and 6.4%
* Physical Activity (less than 150 min/week moderate-intensity Physical Activity, no more than 1 session/week of resistance exercise)

Exclusion Criteria:

* Unstable Cardiovascular Disease
* Uncontrolled hypertension
* Severe hypertriglyceridemia
* History of or active liver disease
* Uncontrolled thyroid disease
* Active cancer diagnosis
* Smoking
* Engaged in exercise or diet program
* History of bariatric surgery
* GI malabsorptive disorders
* Significant diet intolerances
* History of major psychiatric disorder
* presence of alcohol or substance abuse;
* medications affecting weight,
* EI or EE in past 6 months;
* women currently pregnant, lactating, less than 6 months post-partum, or postmenopausal.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Changes in Appetite Rating | Baseline: Pre-Meal , 30 minutes, 60 minutes, 90 minutes, and 120 minutes post meal / Post-intervention(Week 4) :Pre-Meal, 30 minutes, 60 minutes, 90 minutes ,and 120 minutes post meal
  Hunger/Satiety before/after consumption of a meal
Changes in Hormonal Response to Feeding | Baseline: Pre-Meal , 30 minutes, 60 minutes, 90 minutes, and 120 minutes post meal / Post-intervention(Week 4) :Pre-Meal, 30 minutes, 60 minutes, 90 minutes ,and 120 minutes post meal
  Assessment of Ghrelin levels analyzed in blood samples before/after feeding.

SECONDARY OUTCOMES:
Changes in Body Composition | Baseline and Post-intervention(Week 4)
  Measured via BodPod
Changes in Maximal Strength | Baseline and Post-intervention(Week 4)
  Measurement via 10 repetition-max testing.
Changes in Physical Activity Levels | Baseline and Post-intervention(Week 4)
  Measured via ActivPal Monitor
Changes in Food-Related Behaviors | Baseline and Post-intervention(Week 4)
  Evaluated via the Food Craving Inventory
Changes in Food-Related Behaviors | Baseline and Post-intervention(Week 4)
  Evaluated via Three-Factor Eating Questionnaire
Changes in Food-Related Behaviors | Baseline and Post-intervention(Week 4)
  Evaluated via the Weight Efficacy Lifestyle Questionnaire
Change in Ad libitum Energy Intake - In lab | Baseline and Post-intervention(Week 4)
  In lab ad libitum buffet lunch (via weigh and measure methodology)
Changes in Ad libitum Energy Intake - Free Living | Baseline and Post-intervention(Week 4)
  3 days of free-living ad libitum energy intake (via self-report)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya M Halliday, PhD, RD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States